CLINICAL TRIAL: NCT01497366
Title: A Phase 3, Multicenter, Randomized, Active-Controlled Study to Investigate the Safety and Efficacy of PSI-7977 and Ribavirin for 12 Weeks Compared to Pegylated Interferon and Ribavirin for 24 Weeks in Treatment-Naïve Patients With Chronic Genotype 2 or 3 HCV Infection
Brief Title: Phase 3 Study of Sofosbuvir and Ribavirin
Acronym: FISSION
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P7977-1231
Record Dates: First submitted 2011-12-19; First posted 2011-12-22 (Estimated); Results first posted 2014-04-02 (Estimated); Last update posted 2014-04-02 (Estimated); Status verified 2014-03

CONDITIONS: Hepatitis C
Keywords: HCV genotype 2 (GT-2); HCV genotype 3 (GT-3)
MeSH Terms: conditions — Hepatitis C | interventions — Sofosbuvir; peginterferon alfa-2a

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Sofosbuvir+RBV (Experimental): Participants were randomized to receive sofosbuvir+RBV for 12 weeks.
  Interventions: Drug: Sofosbuvir; Drug: RBV
- PEG+RBV (Active Comparator): Participants were randomized to receive PEG+RBV for 24 weeks.
  Interventions: Drug: PEG; Drug: RBV

INTERVENTIONS:
Drug: Sofosbuvir — Sofosbuvir 400 mg (2 × 200 mg tablets) administered orally once daily
  Other Names: Sovaldi™; GS-7977; PSI-7977
  Arms: Sofosbuvir+RBV
Drug: PEG — Pegylated interferon alfa-2a (PEG) 180 μg administered once weekly by subcutaneous injection
  Other Names: Pegasys®
  Arms: PEG+RBV
Drug: RBV — Ribavirin (RBV) administered as 200 mg tablets up to 1200 mg in a divided daily dose
  * Dose of sofosbuvir+RBV group based on baseline weight: < 75kg = 1000 mg and ≥ 75 kg = 1200 mg
  * Dose of PEG+RBV group: 800 mg

SUMMARY:
This study was to assess the safety and efficacy of sofosbuvir (GS-7977; PSI-7977) in combination with ribavirin (RBV) administered for 12 weeks compared with pegylated interferon (PEG)/RBV administered for 24 weeks in treatment-naive patients with Hepatitis C (HCV) genotype 2 or 3. Efficacy was assessed by the rate of sustained viral response (SVR) 12 weeks after the discontinuation of therapy (SVR12). This was a non-inferiority study, and if non-inferiority was demonstrated, the study was then allowed to test for superiority.

ELIGIBILITY:
Inclusion Criteria:

* Chronic Genotype 2 or 3 HCV-infection
* Naive to all HCV antiviral treatment(s)

Exclusion Criteria:

* Positive test at Screening for HBsAg, anti-hepatitis B core immunoglobulin M antibody (anti-HBc IgM Ab), or anti-HIV Ab
* History of any other clinically significant chronic liver disease
* A history consistent with decompensated liver disease
* History or current evidence of psychiatric illness, immunologic disorder, hemoglobinopathy, pulmonary or cardiac disease, seizure disorder or anticonvulsant use, poorly controlled diabetes, cancer, or a history of malignancy, that makes the subject unsuitable for the study.
* Participation in a clinical study within 3 months prior to first dose

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 527 (Actual)
Dates: Start 2011-12; Primary Completion 2013-01 (Actual); Study Completion 2013-04 (Actual)

CONTACTS AND LOCATIONS:
Locations (97):
- United States (67):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Alabama Liver & Digestive Specialist, Montgomery, Alabama
  - Franco Felizarta, MD, Bakersfield, California
  - California Liver Institute, Beverly Hills, California
  - Arrowhead Regional Medical Center, Colton, California
  - SCTI Research Foundation, Coronado, California
  - eStudy Site, La Mesa, California
  - Peter J. Ruane, M.D. Inc., Los Angeles, California
  - eStudySite, Oceanside, California
  - University of California, Davis - Health System, Sacramento, California
  - University of California San Diego Medical Center, San Diego, California
  - Research and Education, Inc., San Diego, California
  - Medical Associates Research Group, Inc., San Diego, California
  - Quest Clinical Research, San Francisco, California
  - South Denver Gastroenterology, PC, Englewood, Colorado
  - Pointe West Infectious Diseases, Bradenton, Florida
  - Midway Immunology & Research Center, LLC, Ft. Pierce, Florida
  - University of Florida College of Medicine, Gainesville, Florida
  - Borland-Groover Clinic Baptist, Jacksonville, Florida
  - University of Miami, School of Medicine, Miami, Florida
  - Orlando Immunology Center, Orlando, Florida
  - Internal Medicine Specialists, Orlando, Florida
  - Advanced Research Institute, Trinity, Florida
  - South Florida Center of Gastroenterology, Wellington, Florida
  - AIDS Research Consortium of Atlanta, Inc., Atlanta, Georgia
  - Atlanta Gastroenterology Associates, Atlanta, Georgia
  - Gastrointestinal Specialists of Georgia, PC, Marietta, Georgia
  - University of Chicago, Chicago, Illinois
  - Indianapolis Gastroenterology Research Foundation, Indianapolis, Indiana
  - Digestive Disease Associates, P.A., Baltimore, Maryland
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - The Research Institute, Springfield, Massachusetts
  - Partners in Internal Medicine, PC, Worcester, Massachusetts
  - University of Massachusetts, Worcester, Worcester, Massachusetts
  - Henry Ford Health System, Detroit, Michigan
  - Digestive Health Specialists, PA, Tupelo, Mississippi
  - Veterans Affairs Medical Center, East Orange, New Jersey
  - AGA Clinical Research Associates, LLC, Egg Harbor, New Jersey
  - ID Care, Hillsborough, New Jersey
  - Atlantic Research Affiliates, LLC, Morristown, New Jersey
  - Southwest C.A.R.E. Center, Santa Fe, New Mexico
  - North Shore University Hospital, Manhasset, New York
  - Weill Cornell Medical College, New York, New York
  - Mount Sinai School of Medicine, New York, New York
  - University of Rochester, Rochester, New York
  - Asheville Gastroenterology Associates, P.A., Asheville, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - Carolinas Center for Liver Disease, Statesville, North Carolina
  - Digestive Health Specialists, PA, Winston-Salem, North Carolina
  - University of Cincinnati, Cincinnati, Ohio
  - Gastroenterology United of Tulsa, Tulsa, Oklahoma
  - Schleinitz Research and Gastroenterology LLC, Medford, Oregon
  - Regional Gastroenterology Associates of Lancaster, Ltd., Lancaster, Pennsylvania
  - UPMC Center For Liver Diseases, Pittsburgh, Pennsylvania
  - University Gastroenterology, Warwick, Rhode Island
  - Gastro One, Germantown, Tennessee
  - Nashville Gastrointestinal Specialists Inc., Nashville, Tennessee
  - Texas Clinical Research Institute, LLC, Arlington, Texas
  - Baylor University Medical Center, Dallas, Texas
  - Kelsey-Seybold Clinic PA, Houston, Texas
  - Research Specialists of Texas, Houston, Texas
  - VAMC & Baylor College, Houston, Texas
  - Alamo Medical Research, San Antonio, Texas
  - Metropolitan Research, Fairfax, Virginia
  - Digestive and Liver Disease Specialist, Ltd., Norfolk, Virginia
  - Digestive and Liver Disease Specialists, Norfolk, Virginia
  - Virginia Mason Medical Center, Seattle, Washington
- Australia (14):
  - Canberra Hospital, Garran, Australian Capital Territory
  - Royal Prince Alfred Hospital, Camperdown, New South Wales
  - Concord Repatriation General Hospital, Concord, New South Wales
  - St. George Hospital, Kogarah, New South Wales
  - Gallipoli MRF, Greenslopes, Queensland
  - Royal Brisbane Hospital Research Foundation, Herston, Queensland
  - Princess Alexandria, Woollongabba, Queensland
  - Royal Adelaide Hospital, Adelaide, South Australia
  - Monash Medical Centre, Clayton, Victoria
  - Austin Hospital, Heidelberg, Victoria
  - The Alfred, Melbourne, Victoria
  - Fremantle Hospital, Fremantle, Western Australia
  - Sir Charles Gairdner, Nedlands, Western Australia
  - Royal Perth Hospital, Perth, Western Australia
- Canada (5):
  - (G.I.R.I.) Gastrointestinal Research Institute, Vancouver, British Columbia
  - Mount Sinai Hospital, Toronto, Ontario
  - University Health Network-Toronto Western Hospital, Toronto, Ontario
  - Toronto Liver Centre, Toronto, Ontario
  - Toronto Digestive Disease Associates, Inc., Vaughan, Ontario
- Casa Sollievo della Sofferenza Hospital, San Giovanni Rotondo, Italy
- Academish Medisch Centrum, Amsterdam, Netherlands
- New Zealand (6):
  - Auckland City Hospital, Grafton, Auckland
  - Tauranga Hospital, Tauranga, BOP
  - Christchurch Hospital, Chrischurch, Canterbury
  - Mercy Hospital, Dunedin, OTA
  - Waikato Hospital (District Health Board), Hamilton, Waikato Region
  - Wellington Hospital, Newtown, WGN
- Fundacion de Investigacion de Diego, San Juan, Puerto Rico, Puerto Rico
- Sweden (2):
  - Sahlgrenska Universitetssjukhuset, Östra Sjukhus, Gothenburg
  - Karolinska Universitetssjukhuset, Solna, Stockholm

REFERENCES:
- [Derived] Stepanova M, Nader F, Cure S, Bourhis F, Hunt S, Younossi ZM. Patients' preferences and health utility assessment with SF-6D and EQ-5D in patients with chronic hepatitis C treated with sofosbuvir regimens. Aliment Pharmacol Ther. 2014 Sep;40(6):676-85. doi: 10.1111/apt.12880. Epub 2014 Jul 15. PMID 25040192
- [Derived] Lawitz E, Mangia A, Wyles D, Rodriguez-Torres M, Hassanein T, Gordon SC, Schultz M, Davis MN, Kayali Z, Reddy KR, Jacobson IM, Kowdley KV, Nyberg L, Subramanian GM, Hyland RH, Arterburn S, Jiang D, McNally J, Brainard D, Symonds WT, McHutchison JG, Sheikh AM, Younossi Z, Gane EJ. Sofosbuvir for previously untreated chronic hepatitis C infection. N Engl J Med. 2013 May 16;368(20):1878-87. doi: 10.1056/NEJMoa1214853. Epub 2013 Apr 23. PMID 23607594

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were enrolled in a total of 90 study sites in the United States, Australia, New Zealand, Canada, Sweden, Italy, and the Netherlands. The first participant was screened on 19 December 2011. The last participant observation was on 08 April 2013.
Pre-assignment Details: 666 participants were screened and 527 were randomized; 499 participants received at least 1 dose of study drug, and comprise the Safety Analysis Set. The 496 participants with genotype 2 or 3 HCV infection who were randomized and received at least 1 dose of study drug comprise the Full Analysis Set.
Groups:
- Sofosbuvir+RBV: Participants were randomized to receive sofosbuvir+ribavirin (RBV) for 12 weeks.
Period: Overall Study
Arm/Group | Sofosbuvir+RBV | PEG+RBV
Started | 263 | 264
Randomized But Not Treated | 7 | 21
Completed | 224 | 176
Not Completed | 39 | 88
Not completed — Virologic failure | 2 | 50
Not completed — Lost to Follow-up | 11 | 10
Not completed — Withdrawal by Subject | 6 | 6
Not completed — Initiated Non-protocol HCV Treatment | 7 | 0
Not completed — Other | 5 | 0
Not completed — Death | 1 | 1
Not completed — Randomized but not treated | 7 | 21

BASELINE CHARACTERISTICS:
Population: Safety Analysis Set
Groups:
- Total: Total of all reporting groups
Arm/Group | Sofosbuvir+RBV | PEG+RBV | Total
Number analyzed (Participants) | 256 | 243 | 499
Age, Continuous [Mean (Standard Deviation); unit: years] | 48 (10.8) | 48 (11.4) | 48 (11.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 85 | 87 | 172
  Male | 171 | 156 | 327
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 41 | 31 | 72
  Not Hispanic or Latino | 215 | 212 | 427
  Unknown or Not Reported | 0 | 0 | 0
Race/Ethnicity, Customized [Number; unit: participants]
  Black or African American | 12 | 5 | 17
  White | 223 | 212 | 435
  Asian | 14 | 15 | 29
  American Indian/Alaska Native/First Nations | 4 | 4 | 8
  Hawaiian or Pacific Islander | 2 | 6 | 8
  Black and White | 1 | 0 | 1
  South American | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  United States | 165 | 151 | 316
  Canada | 15 | 24 | 39
  Australia | 32 | 29 | 61
  Netherlands | 3 | 1 | 4
  Italy | 8 | 4 | 12
  New Zealand | 29 | 30 | 59
  Sweden | 4 | 4 | 8
Hepatitis C Virus (HCV) genotype [Number; unit: participants]
  Genotype 1 | 3 | 0 | 3
  Genotype 2 | 70 | 67 | 137
  Genotype 3 | 183 | 176 | 359
Baseline HCV RNA [Mean (Standard Deviation); unit: log10 IU/mL] | 6.0 (0.82) | 6.0 (0.78) | 6.0 (0.80)
Baseline HCV RNA Category [Number; unit: participants]
  < 6 log10 IU/mL | 108 | 106 | 214
  ≥ 6 log10 IU/mL | 148 | 137 | 285
IL28b genotype [Number; unit: participants]
  CC | 108 | 106 | 214
  CT | 121 | 98 | 219
  TT | 25 | 38 | 63
  Missing | 2 | 1 | 3
Cirrhosis [Number; unit: participants]
  No | 205 | 189 | 394
  Yes | 50 | 50 | 100
  Missing | 1 | 4 | 5

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Sustained Virologic Response 12 Weeks After Stopping All Study Drugs (SVR12)
Description: SVR12 was defined as HCV RNA < the lower limit of quantitation (LLOQ; < 25 IU/mL) 12 weeks after study drug cessation.
Time Frame: Post-treatment Week 12
Population: Full Analysis Set
Measure: Number; unit: percentage of participants
Arm/Group | Sofosbuvir+RBV | PEG+RBV
Number analyzed (Participants) | 253 | 243
percentage of participants | 67 [61.0 to 72.9] | 67 [60.4 to 72.6]
Statistical Analysis 1: Comparison: Sofosbuvir+RBV vs PEG+RBV; Test type: Non-Inferiority or Equivalence — Non-inferiority would be demonstrated if the lower bound of the 2-sided 95% confidence interval (CI) for the difference in SVR12 rates was greater than -15%; Difference in percentages = 0.3, 95% CI 2-sided [-7.5 to 8.0] — The difference in percentages between treatment groups and the 95% CI calculated were based on stratum adjusted Mantel-Haenszel proportions

2. Secondary Outcome: Number of Participants Who Experienced Adverse Events (AEs) and Graded Laboratory Abnormalities
Time Frame: Up to 24 weeks plus 30 days following the last dose of study drug
Population: Safety Analysis Set
Measure: Number; unit: participants
Arm/Group | Sofosbuvir+RBV | PEG+RBV
Number analyzed (Participants) | 256 | 243
participants
  AEs leading to discontinuation of any study drug | 3 | 29
  Serious AEs | 7 | 3
  Grade 3 laboratory abnormalities | 33 | 80
  Grade 4 laboratory abnormalities | 3 | 21
  Deaths | 1 | 0

3. Secondary Outcome: Percentage of Participants With Sustained Virologic Response 24 Weeks After Stopping All Study Drugs (SVR24)
Description: SVR24 was defined as HCV RNA < LLOQ 24 weeks after study drug cessation.
Time Frame: Post-treatment Week 24
Population: Full Analysis Set
Measure: Number; unit: percentage of participants
Arm/Group | Sofosbuvir+RBV | PEG+RBV
Number analyzed (Participants) | 253 | 243
percentage of participants | 66.8 [60.6 to 72.6] | 65.4 [59.1 to 71.4]

4. Secondary Outcome: Percentage of Participants With HCV RNA < LLOQ on Treatment
Time Frame: Up to 12 Weeks
Population: Participants in the Full Analysis Set with available data were analyzed.
Measure: Number; unit: percentage of participants
Groups:
- Sofosbuvir+RBV: Participants were randomized to receive sofosbuvir (SOF)+RBV for 12 weeks.
Arm/Group | Sofosbuvir+RBV | PEG+RBV
Number analyzed (Participants) | 253 | 243
percentage of participants
  Week 1 (SOF+RBV, n = 252; PEG+RBV, n = 243) | 43.7 | 6.6
  Week 2 (SOF+RBV, n = 251; PEG+RBV, n = 241) | 92.0 | 31.5
  Week 4 (SOF+RBV, n = 250; PEG+RBV, n = 236) | 99.6 | 66.9
  Week 8 (SOF+RBV, n = 248; PEG+RBV, n = 231) | 99.6 | 85.7
  Week 12 (SOF+RBV, n = 244; PEG+RBV, n = 224) | 99.2 | 92.4

5. Secondary Outcome: Change From Baseline in HCV RNA
Time Frame: Baseline to Week 12
Population: Participants in the Full Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: log10 IU/mL
Arm/Group | Sofosbuvir+RBV | PEG+RBV
Number analyzed (Participants) | 253 | 243
log10 IU/mL
  Week 1 (SOF+RBV, n = 239; PEG+RBV, n = 236) | -4.26 (0.689) | -2.19 (1.287)
  Week 2 (SOF+RBV, n = 246; PEG+RBV, n = 233) | -4.60 (0.820) | -3.19 (1.572)
  Week 4 (SOF+RBV, n = 250; PEG+RBV, n = 235) | -4.64 (0.816) | -4.04 (1.389)
  Week 8 (SOF+RBV, n = 248; PEG+RBV, n = 228) | -4.63 (0.850) | -4.42 (1.163)
  Week 12 (SOF+RBV, n = 243; PEG+RBV, n = 222) | -4.65 (0.820) | -4.45 (1.226)

6. Secondary Outcome: Percentage of Participants With Virologic Failure During Treatment
Description: Virologic failure was defined as either
  * Viral breakthrough: HCV RNA ≥ 25 IU/mL after having previously had HCV RNA < 25 IU/mL while on treatment, confirmed with 2 consecutive values or last available measurement
  * Viral rebound: > 1 log10 IU/mL increase in HCV RNA from nadir while on treatment, confirmed with 2 consecutive values or last available measurement
  * Non-response: HCV RNA persistently ≥ 25 IU/ml while on treatment (through Week 12)
Time Frame: Baseline up to Week 24
Population: Full Analysis Set
Measure: Number; unit: percentage of participants
Arm/Group | Sofosbuvir+RBV | PEG+RBV
Number analyzed (Participants) | 253 | 243
percentage of participants | 0.4 | 7.4

7. Secondary Outcome: Percentage of Participants With Viral Relapse Following Treatment
Description: Viral relapse was defined as HCV RNA ≥ 25 IU/mL in post-treatment after having achieved < LLOQ at last on-treatment measurement, confirmed with 2 consecutive values or last available measurement.
Time Frame: Up to Post-treatment Week 24
Population: Participants in the Full Analysis Set with available data were analyzed.
Measure: Number; unit: percentage of participants
Arm/Group | Sofosbuvir+RBV | PEG+RBV
Number analyzed (Participants) | 249 | 217
percentage of participants | 30.5 | 22.6

ADVERSE EVENTS:
Time Frame: Up to 24 weeks plus 30 days following the last dose of study drug
Arm/Group | Sofosbuvir+RBV | PEG+RBV
Serious Adverse Events (participants affected / at risk) | 7/256 | 3/243
Other Adverse Events (participants affected / at risk) | 219/256 | 233/243
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Sofosbuvir+RBV (N=256) | PEG+RBV (N=243)
Anaemia (Blood and lymphatic system disorders) | 1 | 0
Atrioventriclar shock (Cardiac disorders) | 0 | 1
Chest pain (General disorders) | 1 | 0
Allergy to arthropod sting (Immune system disorders) | 1 | 0
Cellulitis (Infections and infestations) | 1 | 0
Infection (Infections and infestations) | 0 | 1
Osteomyelitis chronic (Infections and infestations) | 1 | 0
Urinary tract infection (Infections and infestations) | 1 | 0
Clavicle fracture (Injury, poisoning and procedural complications) | 0 | 1
Rib fracture (Injury, poisoning and procedural complications) | 0 | 1
Toxicity to various agents (Injury, poisoning and procedural complications) | 1 | 0
Breast cancer in situ (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Sofosbuvir+RBV (N=256) | PEG+RBV (N=243)
Anaemia (Blood and lymphatic system disorders) | 20 | 28
Neutropenia (Blood and lymphatic system disorders) | 0 | 30
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 23
Nausea (Gastrointestinal disorders) | 46 | 70
Diarrhoea (Gastrointestinal disorders) | 23 | 42
Vomiting (Gastrointestinal disorders) | 17 | 23
Dry mouth (Gastrointestinal disorders) | 10 | 15
Fatigue (General disorders) | 92 | 134
Irritability (General disorders) | 25 | 40
Chills (General disorders) | 7 | 44
Influenza like illness (General disorders) | 7 | 44
Pyrexia (General disorders) | 6 | 33
Pain (General disorders) | 5 | 30
Injection site reaction (General disorders) | 0 | 17
Injection site erythema (General disorders) | 0 | 14
Nasopharyngitis (Infections and infestations) | 13 | 5
Decreased appetite (Metabolism and nutrition disorders) | 17 | 44
Myalgia (Musculoskeletal and connective tissue disorders) | 21 | 40
Arthralgia (Musculoskeletal and connective tissue disorders) | 15 | 35
Back pain (Musculoskeletal and connective tissue disorders) | 9 | 20
Headache (Nervous system disorders) | 64 | 108
Dizziness (Nervous system disorders) | 27 | 33
Insomnia (Psychiatric disorders) | 31 | 71
Depression (Psychiatric disorders) | 14 | 35
Anxiety (Psychiatric disorders) | 11 | 16
Cough (Respiratory, thoracic and mediastinal disorders) | 19 | 21
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 18 | 20
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 14 | 10
Rash (Skin and subcutaneous tissue disorders) | 23 | 43
Pruritus (Skin and subcutaneous tissue disorders) | 19 | 42
Alopecia (Skin and subcutaneous tissue disorders) | 12 | 24
Dry skin (Skin and subcutaneous tissue disorders) | 11 | 23

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
After conclusion of the study and without prior written approval from Gilead, investigators in this study may communicate, orally present, or publish in scientific journals or other media only after the following conditions have been met:

* The results of the study in their entirety have been publicly disclosed by or with the consent of Gilead in an abstract, manuscript, or presentation form; or
* The study has been completed at all study sites for at least 2 years